CLINICAL TRIAL: NCT04802863
Title: A Phase 1, Open-label Study to Evaluate the Safety and Intrapulmonary Pharmacokinetics of XNW4107, Imipenem and Cilastatin in Healthy Subjects
Brief Title: Intrapulmonary Pharmacokinetics of XNW4107, Imipenem and Cilastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: XNW4107-004
Record Dates: First submitted 2021-03-02; First posted 2021-03-17 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Imipenem; Cilastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Five doses of XNW4107 with imipenem/cilastatin (Experimental): Each subject will receive a total of five doses of 250 mg XNW4107 in combination with 500 mg imipenem/500 mg cilastatin via IV infusion administered every 6 hours with each administration infused over 60 minutes.
  Interventions: Drug: XNW4107, Imipenem/Cilastatin

INTERVENTIONS:
Drug: XNW4107, Imipenem/Cilastatin — Five doses of 250 mg XNW4107 in combination with 500 mg imipenem/500 mg cilastatin

SUMMARY:
This is a Phase 1, open-label, single-center study of XNW4107 and imipenem/cilastatin administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

* 1． Adult males or female subjects, between 18 and 55 years of age (both inclusive) at the time of screening;

  2. BMI ≥ 18.5 and ≤ 32 (kg/m²) and weight between 55.0 and 100.0 kg (both inclusive);

  3. Medically healthy without clinically significant abnormalities as assessed by the Investigator based on screening medical history, physical examination, vital signs, 12-lead ECG, hematology, biochemistry, coagulation and urinalysis;

  4. Forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value at screening;

  5. Non-smoker (with no use of other tobacco, nicotine or marijuana-containing products, in any form), as documented by history (no nicotine or marijuana use within 3 months prior to Screening);

  6. Negative urine drug, alcohol or cotinine testing at screening and check-in (Day -1);

  7. Participants of reproductive potential (male or female) must be willing to use contraception

  8. Ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food (coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.) or product containing any of these from 72 hours prior to study drug administration until discharge from the clinical unit.

Exclusion Criteria:

* 1. History or presence of significant oncologic, cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, vascular or neurological disease, including any acute illness or surgery within the past 3 months determined by the Investigator to be clinically relevant;

  2. Recent history (within 6 months) of known or suspected Clostridium difficile infection;

  3. History of seizure disorder;

  4. Positive testing for human immunodeficiency virus antibody (HIV Ab), hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab);

  5. Positive RT-PCR testing for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening;

  6. Close contact with anyone who tested positive for SARS-CoV-2 infection, or presence of symptoms associated with SARS-CoV-2 infection at Screening or Check-in, or within 14 days prior to Screening.

  7. Electrocardiogram (ECG) with QTcF interval duration equal or greater than 450 msec for males and 470 msec for females obtained after at least 5 min in a supine or semi-supine position at quiet rest at Screening or Check-In (Day -1);

  8. Subjects who have any of the following abnormalities on laboratory values at screening or prior confinement including: a. White blood cell count < 3,000/mm³, hemoglobin < 11g/dL; b. Absolute neutrophil count <1,200/mm³, platelet count <120,000/mm³; c. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 1.5 x the upper limit of normal (ULN) for the reference laboratory;

  9. History of substance abuse or alcohol abuse within the previous 5 years;

  10. Use of prescription medications (with the exception of hormone replacement therapy and contraceptives listed in inclusion criterion #10), including nonsteroidal anti-inflammatory drugs, sucralfate, or herbal preparations within 7 days before Check in (Day -1), or use of an over-the-counter medication, acetaminophen (>2 g/day), vitamins, or supplements (including fish liver oils) within 7 days before Check in (Day -1); or probenecid or valproic acid within 30 days before Check in (Day -1);

  11. History of hypersensitivity to β-lactam antibiotics or drugs that include sulfobutylether β-cyclodextrin sodium (SBECD) as an excipient (e.g. Tegretol, Vfend, Geodon and Noxafil);

  12. History of significant multiple and/or severe allergies (including latex allergy); anaphylactic reaction; or significant prescription drug, non-prescription drug, or food intolerance.

  13. Donation of blood or plasma within 30 days prior to Check-In (Day-1), or loss of whole blood of more than 500 mL within 30 days prior to Check-In (Day-1), or receipt of a blood transfusion within 1 year of study enrollment;

  14. Participation in another investigational clinical trial within 30 days prior to screening;

  15. A female who is pregnant or breastfeeding;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Area under the concentration curve (AUC) from time zero to the last quantifiable sample (AUC0-t) of plasma PK and lung penetration of XNW4107, imipenem and cilastatine in healthy adult volunteers. | From baseline to 12 hours post- fifth dose
AUC extrapolated to infinity (AUC0-∞) of plasma PK and lung penetration of XNW4107, imipenem and cilastatin in healthy adult volunteers. | From baseline to 12 hours post- fifth dose
AUC from time zero to 6 hours after start of the infusion (AUC0-6) of plasma PK and lung penetration of XNW4107, imipenem and cilastatin in healthy adult volunteers. | From baseline to 6 hours post- fifth dose
Maximum concentration (Cmax) of plasma PK and lung penetration of XNW4107, imipenem and cilastatin in healthy adult volunteers. | From baseline to 12 hours post- fifth dose
Minimum concentration (Cmin) of plasma PK and lung penetration of XNW4107, imipenem and cilastatin in healthy adult volunteers. | From baseline to 12 hours post- fifth dose
Time to Cmax (tmax) of plasma PK and lung penetration of XNW4107, imipenem and cilastatin in healthy adult volunteers. | From baseline to 12 hours post- fifth dose
The terminal-phase half-life (t1/2) of plasma PK and lung penetration of XNW4107, imipenem and cilastatin in healthy adult volunteers. | From baseline to 12 hours post- fifth dose

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events of Hematology as assessed by CTCAE v5.0 | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Hematology including White cell count with differential (total and % of neutrophil, lymphocyte, monocyte, eosinophil, and basophil), red blood cell count in m/mm³, hemoglobin in g/dL, hematocrit in % and platelet count m/mm³.
Number of participants with treatment-related adverse events of Coagulation as assessed by CTCAE v5.0. | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Coagulation including Prothrombin time in seconds, activated partial thromboplastin time in seconds and International Normalized Ratio (INR).
Number of participants with treatment-related adverse events of Biochemistry as assessed by CTCAE v5.0. | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Biochemistry including Sodium in mmol/L, calcium in mg/dL, phosphate in mg/dL, potassium in mmol/L, chloride in mmol/L, glucose in mg/ dl, BUN in mg/dl, uric acid in mg/dl, creatinine in mg/dL, creatine kinase in IU/L, creatinine clearance calculated in ml/ min/1.73m² , total bilirubin in mg/dL, direct bilirubin in mg/dL, alkaline phosphatase in IU/L, ALT in IU/L, AST in IU/L, lactate dehydrogenase in IU/L, gamma-glutamyl transferase in IU/L, total protein in g/dL, albumin in g/dL, triglycerides in mg/dL, and cholesterol in mg/dL.
Number of participants with treatment-related adverse events of Urinalysis as assessed by CTCAE v5.0. | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in clinical laboratory values of Urinalysis Specific gravity, pH, leukocyte esterase, protein, glucose, ketones, bilirubin, blood, nitrite, urobilinogen. [Time
Number of participants with treatment-related adverse events of Physical Examination as assessed by CTCAE v5.0. | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in Physical Examination of the following body systems: HEENT; cardiovascular, respiratory, gastrointestinal, dermatological, musculoskeletal, nervous systems, lymph nodes and general appearance, and in kilograms, height in meters and weight and height will be combined to report BMI in kg/m².
Number of participants with treatment-related adverse events of Vital Signs as assessed by CTCAE v5.0. | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in Vital Signs (Systolic and diastolic blood pressure in mmHg, heart rate in Beats per min, respiratory rate in Breaths per min, and oral temperature in Degree celsius).
Number of participants with treatment-related adverse events of 12-Lead Electrocardiogram (ECG) as assessed by CTCAE v5.0. | From baseline up to Day 9
  Safety and tolerability up to the last study visit as assessed by the incidence of treatment-emergent AEs along with clinically significant changes from baseline in 12-Lead Electrocardiogram including heart rate(bpm), RR interval(ms), PR interval(ms), QRS(ms), QT(ms) and QTcF(ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Associates PA, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No